CLINICAL TRIAL: NCT01475500
Title: Nashville Early Diagnosis Lung Cancer Project
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Grogan, Associate Professor - Thoracic Surgery, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC THO 1078; U01CA152662 (NIH)
Record Dates: First submitted 2011-10-18; First posted 2011-11-21 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Respiratory Physiological Phenomena; Bronchoscopy; Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, Blood, Urine, Nasal brushings, Buccal cells, Bronchical washings, Bronchioalveolar lavage brushings, Endobronchial biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Screening: These high-risk subjects will undergo screening for lung cancer. All subjects will undergo all listed interventions
  Interventions: Procedure: Sputum sample; Procedure: Pulmonary function tests; Radiation: Computerized tomography (CT) scan of the chest; Other: Buccal epithelium collection; Procedure: Nasal brushings; Procedure: Bronchoscopy; Procedure: Bronchoalveolar lavage; Procedure: Blood sample collection; Procedure: Urine sample; Procedure: Questionnaire-data collection

INTERVENTIONS:
Procedure: Sputum sample — This is a collection of sputum (mucous) you cough up. Three morning samples will be collected at one time. Sputum will be collected at baseline, year 1, year 2 and year 5.
Procedure: Pulmonary function tests — A series of different breathing tests designed to measure lung function and to determine the presence or absence of chronic obstructive pulmonary disease will be performed at baseline.
Radiation: Computerized tomography (CT) scan of the chest — A CT scan uses x-rays to take detailed pictures of the chest. Performed at baseline, year 2 and year 5. If nodules are present, CT scans will be performed every 3 months for the first year of the study.
Other: Buccal epithelium collection — Collect cells from the inside of the cheek. Samples will be collected at baseline and yearly to year 5.
Procedure: Nasal brushings — A cytobrush is used to remove cells on the surface of the inside of the nose. Samples will be collected at baseline and yearly to year 5.
Procedure: Bronchoscopy — A flexible tube with a light and a camera will be inserted through the nose or mouth, and into the lungs to look at the airway. Bronchial tissue will be obtained.
Procedure: Bronchoalveolar lavage — During a bronchoscopy, a flexible tube with a light and a camera is passed through the mouth or nose into the lungs and fluid is squirted into a small part of the lung and collected for examination. Bronchoscopies will be performed at baseline and at year 5.
Procedure: Blood sample collection — A venous blood sample will be collected for testing of biomarkers and other relevant tests. Blood will be taken at baseline and yearly to year 5.
Procedure: Urine sample — Urine will be collected for routine urine tests at baseline and yearly to year 5.
Procedure: Questionnaire-data collection — A questionnaire about the patient's health, medical, and smoking history. Administered at baseline and yearly to year 5. Data will be taken from patient interviews and from the medical record.

SUMMARY:
This screening study will address the lack of molecular strategies for the early detection of lung cancer and integrate those with epidemiological and imaging strategies.

The hypothesis is that the repeated measure of biomarkers of risk obtained from the molecular analysis of biological specimens including those from bronchoscopy (bronchial brushings and biopsies) may contribute to the refinement of high-risk populations and allow an earlier clinical diagnosis.

The goal of the investigators study is to provide screening for lung cancer in a high-risk population. In this prospective cohort it will be tested whether repeated measure of biomarkers of risk allows early detection of lung cancer.

DETAILED DESCRIPTION:
It is proposed to test the hypotheses in a screening study of high risk individuals (characterized by an established prediction rule). The expected prevalence of lung cancer in this high risk group is estimated to be 2% per year. All individuals benefit from clinic visit, low-dose Chest CT, spirometry and auto-fluorescence bronchoscopy at baseline, Chest CT, follow-up doctor visit, and auto-fluorescence bronchoscopy at least at year 2 and 5.

ELIGIBILITY:
Inclusion Criteria:

* 55 - 80 years of age
* Current smoker or former smoker. If former smoker, must have quit smoking less than 15 years ago
* >/= 30 pack year of smoking history

Exclusion Criteria:

* History of diagnosis/treatment of lung cancer in the past 2 years
* History of head/neck or esophageal cancer in the last 1 year
* Inability to provide informed consent
* Participants in whom stopping anti-platelet or anti-coagulation therapy would have an adverse effect (DVT, mechanical heart valves, unstable coronary syndrome, etc.)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: By physician referral, medical professional referral or self-referral
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To compare candidate biomarkers over time among participants who did and did not develop lung cancer | at baseline and yearly to year 5
  Blood, sputum, urine, nasal washings, buccal epithelium, endobronchial tissue, and bronchioalveolar washings are examined for biomarkers present in patients who develop lung cancer compared with those patients who do not develop lung cancer. Baseline and yearly screening results will be compared in the two groups.

SECONDARY OUTCOMES:
To identify and validate new biomarkers that are associated with lung cancer risk factors and premalignant lesions. | at baseline and yearly to year 5
  Blood, sputum, urine, nasal washings, buccal epithelium, endobronchial tissue, and bronchioalveolar washings are examined for presently unknown biomarkers that occur in patients with lung cancer and in patients who do not have lung cancer but who may be at further increased risk of lung cancer.
To assess changes in prevalence and grade of pre-invasive lesions in this cohort. | baseline, at years 2 and 5 (abnormal tissue will re-examined every 6 months)
  Endobronchial tissue will be examined under a microscope for presence of changes in the cells that are abnormal but which are not invasive cancer.
To describe patients eligible for future chemoprevention clinical trials. | at year 5
  Inclusion criteria for those patients who, based on their biomarker profile, are at increased risk of invasive lung cancer and who may benefit from clinical trials that will study chemoprevention strategies for lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grogan, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Veterans Administration, Nashville, Tennessee
  - Vanderbilt University, Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Lakhani DA, Chen SC, Antic S, Muterspaugh A, Cook C, Liu N, Shujat H, Jouan S, Winston B, Fields K, Wenstrup J, Block SL, Hinton A, Miller A, Atmajoana S, Helton JT, Patel K, Balar AB, Brewer K, Nag S, Singh R, Disher A, Huerta L, Fremont R, Rickman O, Chen H, Eisenberg R, Sandler KL, Paulson A, Walker RC, Shah C, Smith GT, Landman B, Deppen S, Grogan EL, Aldrich MC, Massion PP. Establishing a Cohort and a Biorepository to Identify Biomarkers for Early Detection of Lung Cancer: The Nashville Lung Cancer Screening Trial Cohort. Ann Am Thorac Soc. 2021 Jul;18(7):1227-1234. doi: 10.1513/AnnalsATS.202004-344OC. PMID 33400907